CLINICAL TRIAL: NCT07315126
Title: Reliability of Transcutaneous Bilirubin Measurement According to the Skin Colour of Newborns
Acronym: BILICOLOR
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251268; IDRCB (Other: 2025-A01901-48)
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Jaundice
Keywords: Neonatal jaundice; Kernicterus; Newborn
MeSH Terms: conditions — Jaundice, Neonatal; Kernicterus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Single-arm study including 510 patients meeting identical inclusion and exclusion criteria and receiving the same intervention. All participants are enrolled in one study group. Subgroup analyses according to Fitzpatrick skin phototype are planned and are described in the Detailed Description section.
  Interventions: Procedure: Skin color assessment

INTERVENTIONS:
Procedure: Skin color assessment — Each participant's skin color is evaluated according to the Fitzpatrick skin type classification. All other care is standard, and no additional treatment is administered.

SUMMARY:
Neonatal jaundice is a physiological process characterized by a yellow coloration of the skin and mucous membranes linked to an increase in a pigment: bilirubin. However, an excessive accumulation of bilirubin can lead to neurological complications: kernicterus. The screening for pathological jaundice is carried out through daily measurements of transcutaneous bilirubin using non-invasive devices (bilirubinometers). The diagnosis is made by measuring blood bilirubin levels and comparing them with reference curves. In newborns with dark skin, transcutaneous bilirubin measurements may be inaccurate because melanin interferes with the bilirubinometers.

DETAILED DESCRIPTION:
Neonatal jaundice is a physiological process characterized by a yellow coloration of the skin and mucous membranes. It is caused by an accumulation of bilirubin in the blood. Bilirubin is a product of haemolysis, the breakdown of haem. It circulates in the blood bound to albumin. The unconjugated fraction that is not bound to albumin is neurotoxic. This physiological process must be monitored because free bilirubin is neurotoxic. Due to the immaturity of the blood-brain barrier, it can cross into the brain and damage the basal ganglia. In this case, the condition is referred to as kernicterus, which can cause acute and then chronic encephalopathies, leading to neurosensory disorders and disability in children.

Prevention of kernicterus relies on the detection of excessively high bilirubin concentrations. However, diagnosis requires an invasive blood sample to measure serum bilirubin level. Clinical screening based on the color of the newborn's skin and eyes is insufficient and must be complemented by non-invasive photometric screening using a transcutaneous bilirubinometer (a light flash on the skin). The device estimates the level of bilirubin in the blood. Measurements are performed daily by midwives during the mother and newborn's stay in the maternity ward within the first 3 to 5 days after birth. Unfortunately, the reliability of this screening appears to be lower in newborns with darker skin tones.

Between 2011 and 2012, the National Reference Center for Perinatal Hemobiology (CNRHP) recorded five cases of kernicterus in France, two of which involved delayed screening due to the newborns' dark skin. In both cases, an exchange transfusion (the last-resort treatment) had to be performed. In 2019, N'Guessan et al. reported a similar case in which, despite the presence of jaundice risk factors and a transcutaneous bilirubin level above the alert threshold, the medical team was reassured and concluded that the high reading was a discrepancy related to the infant's dark skin, without performing a confirmatory blood test.

Although most studies show a good correlation between transcutaneous bilirubin (TcB) and serum bilirubin (TSB) levels, they all report an overestimation of TcB values in newborns with darker skin. This does not generally compromise the detection of severe jaundice but may lead to a greater number of invasive blood samples to verify the results.

The methodology of most of these studies is questionable, as they refer to older-generation photometric devices, or use unvalidated colorimetric scales, and sometimes even subjective clinical assessments to determine skin color.

In 2017, a study including 6,373 preterm African-American newborns proposed a specific transcutaneous bilirubin nomogram for dark-skinned infants, with adjusted thresholds for BiliCheck© and JM-103© devices. However, these specific curves have never been externally validated and are therefore not used in routine clinical practice.

The question of the reliability of transcutaneous bilirubin measurements for jaundice screening according to skin color thus remains highly relevant.

To increase knowledge on the subject, it seems necessary to us to carry out a rigorous study of the reliability of transcutaneous bilirubin measurements performed routinely with a new-generation bilirubinometer for the screening of jaundice according to skin color. The children will be classified into three skin color groups using the Fitzpatrick classification: light skin, intermediate skin, and dark skin.

ELIGIBILITY:
Inclusion Criteria:

* Born from 36 weeks of amenorrhea
* Hospitalized in the postnatal ward or kangaroo care unit
* Requiring a blood test for bilirubin analysed at the Cochin laboratory.
* No objection from both holders of parental authority.

Exclusion Criteria:

* Having received phototherapy treatment within the last 24 hours

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns from 36 weeks of amenorrhea hospitalized in the postnatal ward or in the kangaroo unit within the Port-Royal maternity.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the reliability of transcutaneous bilirubin measurements performed routinely with a new-generation bilirubinometer to screen for jaundice according to the degree of skin pigmentation of newborns, determined using a published scale, the Fitzpa | First two days of life
  Based on the first transcutaneous and serum bilirubin assessments

SECONDARY OUTCOMES:
To evaluate whether the reliability of transcutaneous bilirubin measurements differs between newborns with dark or intermediate skin phototypes and those with light skin phototyp | 1 to 7 days
  Correlation coefficients between transcutaneous bilirubin and serum bilirubin in the three skin pigmentation groups (light, intermediate, dark)
To compare transcutaneous and serum bilirubin values within each skin pigmentation group and across the overall population | First two days of life
  First measurement of transcutaneous and serum bilirubin performed during newborn follow-up
To estimate the probability that a positive screening result truly corresponds to jaundice in the newborn, according to the degree of skin pigmentation and in the overall population | 1 to 7 days
  Positive predictive value (PPV) of the current screening method-based on a common nomogram for all newborns and jaundice risk factors-according to skin pigmentation level and in the overall population
To determine, according to the degree of skin pigmentation and in the overall population, the number of invasive blood samples performed due to an overestimation of transcutaneous bilirubin when serum bilirubin levels were within physiological ranges | 1 to 7 days
  Rate of invasive blood samples performed in newborns with physiological serum bilirubin levels, according to skin pigmentation level and in the overall population
To determine, in newborns with intermediate or dark phototypes, based on the specific nomograms published in 2017 and integrated into the screening algorithm, the number of invasive blood samples avoided, and to specify whether these cases actually corre | 1 to 7 days
  Rate of invasive samples avoided in newborns with intermediate/dark phototypes thanks to the use of the specific curves published in 2017 (bilirubinometer JM-103) integrated into the screening algorithm, distinguishing cases with or without jaundice
To describe the evolution of the newborns' phototype during the first days of life and assess its potential impact on the reliability of transcutaneous bilirubin measurements | 1 to 7 days
  Fitzpatrick scale and measurements of transcutaneous and serum bilirubin during newborn follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Maternité Port Royal, Paris, France

IPD SHARING:
Plan to Share IPD: No